CLINICAL TRIAL: NCT03941912
Title: An Evaluation of the Erchonia EVRL on Neck and Shoulder Pain of Musculoskeletal Origin
Brief Title: The Effect of Low Level Laser Therapy on Neck and Shoulder Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Erchonia Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: EVRL
Record Dates: First submitted 2019-05-06; First posted 2019-05-08 (Actual); Results first posted 2021-10-14 (Actual); Last update posted 2021-10-14 (Actual); Status verified 2021-10

CONDITIONS: Musculoskeletal Pain
MeSH Terms: conditions — Musculoskeletal Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Erchonia EVRL (Experimental): 635 nanometers (nm) and 405 nm dual-diode laser application
  Interventions: Device: Erchonia EVRL

INTERVENTIONS:
Device: Erchonia EVRL — Single treatment with the Erchonia EVRL to the neck and shoulders. The treatment applies 635 nanometers (nm) red diode light and 405 nm violet diode light simultaneously.

SUMMARY:
This study is to see if applying red and violet low level laser light to the neck and shoulders can help to reduce pain in the neck and shoulders.

DETAILED DESCRIPTION:
It is the goal of the current study to demonstrate non-inferiority in efficacy of the Erchonia® EVRL when used in simultaneous dual diode mode (both the red (640 nano-meter (nm)) and violet (405 nm) diodes activated simultaneously) compared to its use with the red diode only activated, for adjunctive use in providing temporary relief of minor chronic neck and shoulder pain of musculoskeletal origin.

ELIGIBILITY:
Inclusion Criteria:

* Subject presents with one or more of chronic neck or shoulder pain.
* Subject is diagnosed with of one or more of osteoarthritis, chronic muscle spasms or cervical and thoracic spine sprain strain.
* Pain is chronic, having persisted for longer than the past 30 days
* Self-reported Pain rating on the 0-100 Visual Analog Scale (VAS) of 50 or greater.
* Willing and able to refrain from consuming any over-the-counter and/or prescription medication(s) and/or herbal supplements intended for the relief of pain and/or inflammation, including muscle relaxants throughout the course of study participation.
* Willing and able to refrain from engaging in any non-study procedure therapies throughout the course of study participation, including conventional therapies such as physical therapy, occupational therapy and hot or cold packs, as well as alternative therapies such as chiropractic care and acupuncture
* 18 years of age or older

Exclusion Criteria:

* Current active chronic pain disease: such as chronic fatigue syndrome and fibromyalgia
* Use of analgesics or muscle relaxants within 7 days prior to study procedure administration.
* Use of systemic corticosteroid therapy (inhaled and topical corticosteroids permitted), narcotics or Botulinum toxin (Botox®) injection in the neck/shoulder region within 30 days prior to study procedure administration.
* Active cancer or treatment for cancer within the last 6 months.
* Unstable cardiac disease, such as recent cardiac arrhythmia, congestive heart failure or myocardial infarction.
* Prior surgery to the neck/shoulder region.
* Known herniated disc injury.
* Active infection, would or other external trauma to the areas to be treated with the laser Medical, physical or other contraindications for or sensitivity to light therapy.
* Serious known mental health illness such as dementia or schizophrenia; psychiatric hospitalization in the past two years.
* Pregnant or breast feeding.
* Participation in a research study within the past 30 days.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2018-04-16 (Actual); Primary Completion 2019-03-10 (Actual); Study Completion 2019-03-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert Silverman, DC, Principal Investigator — Test Site
Locations (2):
- United States (2):
  - Comey Chiropractic Clinic, Largo, Florida
  - New York ChiroCare, White Plains, New York

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Erchonia EVRL
Started | 44
Completed | 44
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Erchonia EVRL
Number analyzed (Participants) | 44
Age, Continuous [Mean (Standard Deviation); unit: years] | 54.07 (14.31)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 27
  Male | 17
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 2
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 38
  More than one race | 0
  Unknown or Not Reported | 3
Region of Enrollment [Number; unit: participants]
  United States | 44
Duration of Neck and Shoulder Pain [Mean (Standard Deviation); unit: months] | 76.58 (110.82)

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Subjects With 30% or Greater Change in Pain Rating on the Visual Analog Scale (VAS)
Description: The Visual Analog Scale (VAS) from one day, baseline to endpoint measurement (following 13-minute treatment administration) is calculated for each subject. Individual subject success is defined as a 30% or greater change in VAS pain scores across the evaluation period. A negative (-) percent change indicates a decrease in pain level and is positive for individual subject success. A positive (+) percent change indicates an increase in pain level and is negative for individual subject success.
  Overall study success criteria is defined as at least 65%±5% (percentage of subjects) meeting the study individual success criteria.
Time Frame: one day
Measure: Number; unit: percentage of subjects
Arm/Group | Erchonia EVRL
Number analyzed (Participants) | 44
percentage of subjects | 75

ADVERSE EVENTS:
Time Frame: 48 hours
Arm/Group | Erchonia EVRL
All-Cause Mortality (participants affected / at risk) | 0/44
Serious Adverse Events (participants affected / at risk) | 0/44
Other Adverse Events (participants affected / at risk) | 0/44

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form: Study Protocol (2018-03-21): https://cdn.clinicaltrials.gov/large-docs/12/NCT03941912/Prot_SAP_ICF_000.pdf